CLINICAL TRIAL: NCT01518179
Title: The Effect of Wearing Made-to-Measure Compression Gloves on Rehabilitation Following DRF.
Brief Title: Compression Gloves for Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Uzi Milman, Director, clinical research unit, Clalit Health Services, Haifa, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-11-0131-CTIL
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Distal Radius Fractures; Fracture of Lower End of Radius; Colles' Fracture; Smith's Fracture
Keywords: Colles' Fracture; Compression Bandages; Occupational therapy; Rehabilitation; Smith's fracture
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Made-to-Measure Compression Gloves (Experimental): Made-to-Measure Compression Gloves in addition to routine follow up and treatment.
  Interventions: Device: Made-to-Measure Compression Gloves
- Control (Other): Routine follow up and treatment
  Interventions: Other: Routine follow up and treatment

INTERVENTIONS:
Device: Made-to-Measure Compression Gloves — Made-to-Measure Compression Gloves in addition to routine follow up and treatment.
  Arms: Made-to-Measure Compression Gloves
Other: Routine follow up and treatment — Control
  Arms: Control

SUMMARY:
Distal Radius Fractures are among the most common orthopedic injuries. Rehabilitation may be characterized by pain, stiffness, swelling, and decreased range of motion (hand and fingers), and grip strength.

Compression gloves are used to enhance rehabilitation after various clinical conditions and injuries. However, there are no reports on the effect of compression gloves following Distal Radius Fracture (DRF).

This study aims to assess the incremental effect of wearing Made-to-Measure Compression Gloves on rehabilitation following DRF.

Working Hypothesis: The addition of Made-to-Measure Compression Gloves to routine follow up and treatment will enhance rehabilitation, when compared with routine follow up and treatment, in patients following Distal Radius Fracture.

ICD 10, Version 2010, conditions to be included in the study (defined jointly as Distal Radius Fractures):

S52.5 Fracture of lower end of radius (Colles' fracture, Smith's fracture) S52.6 Fracture of lower end of both ulna and radius S52.7 Multiple fractures of forearm Excl.: fractures of both ulna and radius: lower end (S52.6), shafts (S52.4).

S52.8 Fracture of other parts of forearm (Lower end of ulna, Head of ulna)

DETAILED DESCRIPTION:
Individuals referred for rehabilitation following DRF will be invited to participate in the study. After obtaining an informed consent individuals will be randomized to receive routine follow up and treatment with or without compression glove. Individuals randomized to made to measure compression gloves will receive them within a week of enrolment. All participating individuals will be assessed by an occupational therapist at enrolment and 2, 4, and 8 week after enrolment. Additional telephone interview, to assess long term effect, will be conducted at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. 4-6 weeks following either surgical or conservative treatment for distal Radius fractures, with or without the involvement of the Ulna.
2. Patients who demonstrate at enrolment at least two of the following:

   * Pain,
   * limited range of motion of the fingers and the wrist,
   * limited strength (weakness of the hand/fingers),
   * swelling /edema,
   * Limited hand functions during performance of Activities of Daily Living (ADL).

Exclusion Criteria:

* Neuropathy
* Peripheral vascular disease
* End stage renal disease
* Previous impairment of fingers/wrist range of motion.
* Previous Lymphedema of the injured hand
* Receiving any additional treatments which is not included in the routine follow up and treatment (i.e. acupuncture, steroids).
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Activities of Daily Living (ADL) by self reported assessment using the Patient Rating Wrist Evaluation (PRWE). | 1 year
  Functional Activities of Daily Living (ADL) by self reported assessment using the Patient Rating Wrist Evaluation (PRWE).

SECONDARY OUTCOMES:
Swelling of the hand and fingers (using CM ribbon) | 10 week
  Swelling of the hand and fingers (using CM ribbon)
Range of motion of the fingers and wrist (using Goniomater) | 10 weeks
  Range of motion of the fingers and wrist (using Goniomater)
Strength of the hand (using the Gamar Dynamometer in KG). | 10 weeks
  Strength of the hand (using the Gamar Dynamometer in KG).
Pain (using VAS as part of PRWE) | 10 weeks
  Pain (using VAS as part of PRWE)
Overall satisfaction of using the compression gloves (using self reported questionnaire). | 10 weeks
  Overall satisfaction of using the compression gloves (using self reported questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Benny Brnfeld, MD, Principal Investigator — Clalit Health Services; Uzi Milman, MD, Study Director — Clalit Health Services; Naomi Schreuer, Ph.D., OTR, Study Chair — Faculty of Social Welfare & Health Sciences, University of Haifa, Haifa, ISRAEL; Inbar Miler, OCT, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Clalit Health Services, Haifa and Western Galilee District, Haifa
  - Clalit Health Services, Haifa

REFERENCES:
- [Result] Miller-Shahabar I, Schreuer N, Katsevman H, Bernfeld B, Cons A, Raisman Y, Milman U. Efficacy of Compression Gloves in the Rehabilitation of Distal Radius Fractures: Randomized Controlled Study. Am J Phys Med Rehabil. 2018 Dec;97(12):904-910. doi: 10.1097/PHM.0000000000000998. PMID 29994792